CLINICAL TRIAL: NCT04313491
Title: Effectiveness of Yoga@Work to Reduce Head and Muscle Pain in Office Workers: Quasi Experimental Study
Brief Title: Effectiveness of Yoga@Work to Reduce Head and Muscle Pain in Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: Brunel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU04
Record Dates: First submitted 2020-03-17; First posted 2020-03-18 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Headache; Cervical Pain; Musculoskeletal Pain
MeSH Terms: conditions — Headache; Neck Pain; Musculoskeletal Pain | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga@Work (Experimental)
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Relaxation yoga exercises, yoga breathing, yoga sound and imagery practices

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of a workplace yoga intervention in reducing the frequency of pain involving the head and neck area.

ELIGIBILITY:
Inclusion Criteria:

* Office workers
* Willing to participate an give consent

Exclusion Criteria:

* Secondary headache
* Neck injury
* Trauma
* Critically ill
* Cognitive impairment
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Frequency of headache, neck and shoulder pain | From baseline to 6-week post intervention
  Pain Journal assessed the number of days with headache, neck and shoulder pain

SECONDARY OUTCOMES:
Severity of head, neck and shoulder pain | From baseline to 6-week post intervention
  Visual Analogue Scale was used to assess the severity of pain with 0 to 10 scale; 0 describe no pain and 10 worst pain.
Analgesics use | From baseline to 6-week post intervention
  Daily pain journal was used to assess analgesics use

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Aarogyam UK; Jaydeep Joshi, BAMS, Study Director — Aarogyam UK; Monomita Nandy, Study Chair — Brunel University
Locations (1):
- Yog Kulam, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided